CLINICAL TRIAL: NCT06269744
Title: A Randomized, Multi-site Trial to Boost Colorectal Cancer Screening Rates Through Proactive Outreach and Navigation in Federally Qualified Health Centers in Brooklyn
Brief Title: Proactive Outreach With FIT
Acronym: PROOF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-01032
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive Screening Outreach (Experimental): Participants assigned to the interventional arm will receive proactive outreach of mailed Fecal Immunochemical Tests (FIT) to screen for colorectal cancer.
  Interventions: Behavioral: Proactive Screening Outreach
- Standard of Care (No Intervention): Participants assigned to the standard of care group will receive usual care (i.e., opportunistic screening for colorectal cancer).

INTERVENTIONS:
Behavioral: Proactive Screening Outreach — Individuals in the interventional arm will receive an information letter, followed by mailed FIT kit. Individuals that do not respond will receive reminder phone calls. Individuals that do respond will receive navigation to assist with completion of FIT and the colonoscopy if FIT is abnormal. Clinic processes will be closely followed and the primary care provider will be informed of the program.
  Arms: Proactive Screening Outreach

SUMMARY:
The purpose of the study is to boost colorectal cancer (CRC) screening rates in an underserved population in Brooklyn through organized, proactive outreach of mailed Fecal Immunochemical Tests (FIT), utilizing evidence-based interventions tailored to the needs of the population.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Men and women aged 45-75
* Receiving medical care at NYULH Flatbush FHC and CHN Crown Heights, East New York, East New York Health Hub, Williamsburg clinic sites.
* Due or overdue for CRC screening.
* Medical visit of any type at clinic in past year.

Providers

* Physicians or primary care givers at Flatbush FHC or CHN Crown Heights, East New York, East New York Health Hub, Williamsburg clinic sites (CHN employees)
* Provide care to CRC screen-eligible patients

Exclusion Criteria:

* Age younger than 45 years old or greater than 75 years old
* Up-to-date with colorectal cancer screening:
* History of colorectal cancer, inflammatory bowel disease, colorectal polyps, or total colectomy
* In hospice care
* Patients 66 years or older living long-term in an institution or with advanced illness
* No address or phone number on file

Providers

• No longer employed at an included clinic site

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants who Complete FIT Test by Month 6 | Up to Month 6

SECONDARY OUTCOMES:
Proportion of Participants with Positive FIT who Complete Colonoscopy by Month 6 | Up to Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Aasma Shaukat, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, Brooklyn, New York
  - Community Health Care Network of New York, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Aasma.Shaukat@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Aasma.Shaukat@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.